CLINICAL TRIAL: NCT06472791
Title: Effect of Centella Asiatica on Vascular Endothelial Function in Older Adults
Brief Title: Centella Asiatica in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Benjamin Zimmerman, Post-Doctoral Research Investigator, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BZCA
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Centella asiatica extract

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to take either a placebo or a Centella Asiatica-containing dietary supplement for four weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Centlla Asiatica (Experimental): 250 mg/day (1 capsules) for week 1. 500 mg/day (2 capsules) for week 2. 750 mg/day (3 capsules) for week 3. 1000 mg/ day (4 capsules) for week 4.
  Interventions: Dietary Supplement: Centella Asiatica
- Placebo (Placebo Comparator): Matched number of capsules per week. Capsules will contain microcrystalline cellulose.
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Centella Asiatica — Centella Asiatica is a perennial, herbaceous plant that is sold as a dietary supplement in the United States under the name Gotu Kola. It has been used for centuries in Ayurvedic and Chinese medicine. Evidence suggests it may help with resilience to aging and cognitive decline. The product for this study will be produced by Arjuna Natural.
  Other Names: gotu kola
  Arms: Centlla Asiatica
Dietary Supplement: Placebo Comparator — The comparator will contain microcystalline cellulose in matched capsules. The comparator product for this study will be produced by Arjuna Natural.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of a dietary supplement containing centella asiatica on on vascular endothelial function in older adults.

ELIGIBILITY:
Inclusion Criteria:

● Age 50 through 85, male or female

* Sufficient proficiency in English to understand study purpose and directions
* Willing and able to give informed consent
* Able to follow protocol and attend visits

Exclusion Criteria:

* History of myocardial infarction, known coronary or carotid disease, or heart failure
* History of stroke, Parkinson's disease, dementia, or other major CNS disorders
* History of hepatic disease (e.g. hepatitis, cirrhosis)
* Recent/recurring history of severe life-threatening medical conditions (e.g. cancer, except non-melanoma skin cancers)
* Active major infectious disease (e.g. pneumonia)
* Heavy alcohol use (15 drinks or more per week for men or 8 drinks or more per week for women) or substance use disorder
* Current use of any medication typically used to treat hypertension or lower blood pressure (e.g. beta-blockers, ACE inhibitors)
* Current use of any medication typically used to prevent the coagulation of blood (e.g. warfarin (Coumadin))
* Chronic NSAID use (>3 times a week for more than 3 months)
* Current use of any medication or supplement typically used as a sedative (e.g. zolpidem (Ambien), benzodiazepines (Valium, Xanax), valerian root)
* Dietary supplements for improving nitric-oxide synthesis (e.g. L-arginine, L-citrulline)
* Current use of any medication typically used to control hypoglycemia (e.g. biguanides (Metformin))
* Current use of any medication typically used for erectile dysfunction (e.g. sildenafil (Viagra), tadalafil (Cialis))
* Pregnant, nursing, or planning a pregnancy within the next 6 weeks
* Open skin rashes and sores that may interfere with the placement of sensors

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial Function | Baseline
  Measured via EndoPAT device through a reactive hyperemia index (RHI).The device measures a signal based on arterial pulsatile volume changes from the fingertip. Blood flow to the brachial artery is temporarily occluded for 5 minutes using a blood pressure cuff. When the pressure is released, the arterial diameter increases, leading to increased flow. The EndoPat software calculates RHI using well-validated methods, by normalizing post-to-pre-occlusion signal ratio in the occluded arm to the same ratio in the control arm. The differences in endothelial function will be measured within groups from Baseline to Week 4. The between group differences will also be analyzed.
Endothelial Function | Day 1
  Measured via EndoPAT device through a reactive hyperemia index (RHI).The device measures a signal based on arterial pulsatile volume changes from the fingertip. Blood flow to the brachial artery is temporarily occluded for 5 minutes using a blood pressure cuff. When the pressure is released, the arterial diameter increases, leading to increased flow. The EndoPat software calculates RHI using well-validated methods, by normalizing post-to-pre-occlusion signal ratio in the occluded arm to the same ratio in the control arm. The differences in endothelial function will be measured within groups from Baseline to Week 4. The between group differences will also be analyzed.
Endothelial Function | Week 4
  Measured via EndoPAT device through a reactive hyperemia index (RHI).The device measures a signal based on arterial pulsatile volume changes from the fingertip. Blood flow to the brachial artery is temporarily occluded for 5 minutes using a blood pressure cuff. When the pressure is released, the arterial diameter increases, leading to increased flow. The EndoPat software calculates RHI using well-validated methods, by normalizing post-to-pre-occlusion signal ratio in the occluded arm to the same ratio in the control arm. The differences in endothelial function will be measured within groups from Baseline to Week 4. The between group differences will also be analyzed.

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | Baseline
  HRV will be measured continually at each visit via a wearable, wireless BodyGuard2.
Heart Rate Variability (HRV) | Day 1
  HRV will be measured continually at each visit via a wearable, wireless BodyGuard2.
Heart Rate Variability (HRV) | Week 4
  HRV will be measured continually at each visit via a wearable, wireless BodyGuard2.
Blood Pressure | Baseline
  Blood pressure will be measured at each visit with an automatic sphygmomanometer.
Blood Pressure | Day 1
  Blood pressure will be measured at each visit with an automatic sphygmomanometer.
Blood Pressure | Week 4
  Blood pressure will be measured at each visit with an automatic sphygmomanometer.
Body Mass Index (BMI) | Baseline
  BMI will be calculated each visit by measuring the participant's height and weight.
Body Mass Index (BMI) | Day 1
  BMI will be calculated each visit by measuring the participant's height and weight.
Body Mass Index (BMI) | Week 4
  BMI will be calculated each visit by measuring the participant's height and weight.

OTHER OUTCOMES:
Adherence | Week 4
  Plasma concentrations of Asiatic Acid
Adherence | Week 4
  Plasma concentrations of Medecassic Acid
Blood glucose | Baseline
  Blood concentrations of glucose
Blood glucose | Week 4
  Blood concentrations of glucose
Urea Nitrogen | Baseline
  Blood concentrations of Urea Nitrogen
Urea Nitrogen | Week 4
  Blood concentrations of Urea Nitrogen
Creatinine | Baseline
  Blood concentrations of creatinine
Creatinine | Week 4
  Blood concentrations of creatinine
Urea Nitrogen to creatinine ratio | baseline
  ratio of blood concentrations of urea nitrogen to creatinine
Urea Nitrogen to creatinine ratio | Week 4
  ratio of blood concentrations of urea nitrogen to creatinine
Sodium | Baseline
  blood concentrations of Sodium
Sodium | Week 4
  blood concentrations of Sodium
Potassium | Baseline
  blood concentrations of Potassium
Potassium | Week 4
  blood concentrations of Potassium
Chloride | Baseline
  blood concentrations of Chloride
Chloride | Week 4
  blood concentrations of Chloride
Carbon Dioxide | baseline
  blood concentration of carbon dioxide
Carbon Dioxide | week 4
  blood concentration of carbon dioxide
Calcium | Baseline
  blood concentration of calcium
Calcium | Week 4
  blood concentration of calcium
Total Protein | Baseline
  Total protein in blood
Total Protein | Week 4
  Total protein in blood
Albumin | Baseline
  Concentration of albumin in blood
Albumin | Week 4
  Concentration of albumin in blood
Globulin | baseline
  Concentration of globulin in blood
Globulin | Week 4
  Concentration of globulin in blood
Albumin to Globulin ratio | Baseline
  Ratio of the blood concentrations of albumin to globulin
Albumin to Globulin ratio | Week 4
  Ratio of the blood concentrations of albumin to globulin
Bilirubin | baseline
  Concentrations of bilirubin in blood
Bilirubin | Week 4
  Concentrations of bilirubin in blood
Alkaline Phosphatase | baseline
  Concentrations of alkaline phosphatase in blood
Alkaline Phosphatase | Week 4
  Concentrations of alkaline phosphatase in blood
aspartate aminotransferase | Baseline
  Concentrations of aspartate aminotransferase in blood
aspartate aminotransferase | Week 4
  Concentrations of aspartate aminotransferase in blood
Alanine aminotransferase | baseline
  Concentrations of Alanine aminotransferase in blood
Alanine aminotransferase | Week 4
  Concentrations of Alanine aminotransferase in blood
Estimated glomerular filtration rate | baseline
  glomerular filtration rate per 1.73 sqM estimated
Estimated glomerular filtration rate | Week 4
  glomerular filtration rate per 1.73 sqM estimated

CONTACTS AND LOCATIONS:
Locations (1):
- Helfgott Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No